CLINICAL TRIAL: NCT02426008
Title: Growth Factors Supplementation to Single-Step Culture Medium
Brief Title: Improving Embryogenesis by Adding Growth Factors to In Vitro Human Culture Media
Acronym: GFSSSCM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ibn Sina Hospital (Other Government)
Collaborators: Banon IVF Center Assiut, Egypt (Other)
Responsible Party: Principal Investigator, Muhammad Fawzy, IVF Lab Director, Ibn Sina Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: IbnSina IVF
Record Dates: First submitted 2015-04-17; First posted 2015-04-24 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: In Vitro Human Embryo Development
MeSH Terms: interventions — Intercellular Signaling Peptides and Proteins

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Culture media with growth factors and Cytokine (Experimental): Growth factors and Cytokine adding to culture media to detect the deference and monitor the embryological outcome.
  Interventions: Other: Growth Factors and Cytokine adding to embryo culture media
- In Vitro culture media (Placebo Comparator): culture media to monitor the embryological outcome as control group
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: Growth Factors and Cytokine adding to embryo culture media
  Arms: Culture media with growth factors and Cytokine
Other: No Intervention — Nothing to Add
  Arms: In Vitro culture media

SUMMARY:
The investigators suppose that adding growth factors that had been found in the female tubal fluid and uterus to In Vitro single step culture media for human embryos might improve the the embryogenesis In Vitro and the clinical outcome of the resulting off spring.

DETAILED DESCRIPTION:
The IVF culture media design and upgrade underwent many ideas during the last 3 decades, we suppose that adding growth factors ( Insulin-like growth factor I, Insulin-like growth factor II, transforming growth factor-beta and epidermal growth factor ) as a promoting growth factors to Lifeglobal culture media might improve embryo development in vitro so we decide to design a trial to compare the embryogenesis by sibling Oocytes of the same patient between to arm of the same culture media and the same culture condition but with one arm with growth factors and the other is traditional one and closely monitor the outcome within the 2 arms and record the results.

ELIGIBILITY:
Inclusion Criteria:

* all patients

Exclusion Criteria:

* over 40 years old

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 426 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Clinical Pregnancy rate ( % ) | 3 months

SECONDARY OUTCOMES:
ongoing Pregnancy rate ( % ) | 6 months
rates of blastocyst formation and quality | 6 days of culture

CONTACTS AND LOCATIONS:
Locations (1):
- Ibnsina IVF center, Sohag, Egypt